CLINICAL TRIAL: NCT00597376
Title: A Six-month, Double-blind, Placebo-controlled, Single Site Study of Cerefolin NAC on Blood Homocysteine, Oxidative Stress, and Beta-amyloid Biomarkers That May Potentiate Inflammation and Neuronal Damage in Older Individuals With Memory Complaints Who Have Not Been Clinically Diagnosed With Mild Cognitive Impairment, Vascular Dementia, or Alzheimer's Disease
Brief Title: Study of the Effects of Cerefolin NAC on Inflammation Blood Markers in Older Individuals With Memory Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Pamlab, Inc. (Industry)
Responsible Party: Principal Investigator, Raj C Shah, Assistant Professor, Family Medicine and Rush Alzheimer's Disease Center, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pamlab-Cerefolin NAC-001-01
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Subjective Memory Loss in Older Persons
Keywords: memory loss
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): On Cerefolin NAC and open-label multivitamin supplement
  Interventions: Other: Cerefolin NAC (a medical food)
- 2 (Placebo Comparator): On placebo and open label multivitamin supplement
  Interventions: Other: Cerefolin NAC placebo

INTERVENTIONS:
Other: Cerefolin NAC (a medical food) — Cerefolin NAC one tablet each day
  Arms: 1
Other: Cerefolin NAC placebo — Placebo tablet once a day
  Arms: 2

SUMMARY:
The purpose of this six-month research study is to determine if Cerefolin NAC reduces levels of substances in the blood that may be associated with thinking ability and the health of brain cells in subjects with memory concerns when compared to a standard multivitamin. Cerefolin NAC is available as a dietary supplement via a prescription from a physician. The multivitamin used in the study contains the Recommended Daily Intake recommended for older persons.

DETAILED DESCRIPTION:
Study Phase: Exploratory

Indication: Memory Complaints

Study Design:

A single-center, double-blind, placebo-controlled study with 100 subjects with memory complaints followed for 6 months (4 visits)using Cerefolin® NAC or placebo once a day in addition to a standardized multivitamin.

Sample Size:

100 subjects as follows:

1. 50 on Cerefolin® NAC + multivitamin; and,
2. 50 on Placebo + multivitamin.

Primary Objective:

To determine if Cerefolin® NAC (compared to multivitamin) decreases the blood level of homocysteine, increases the blood level of glutathione (a marker for oxidative stress), and increases the ratio of Aβ42 to Aβ40 (a marker for beta-amyloid) that may be related to neuronal injury and inflammation.

Secondary Objectives:

1. To determine if Cerefolin® NAC reduces hs-CRP and TNF-α blood levels, and increases IL-6 blood levels.
2. To determine if Cerefolin® NAC (compared to Placebo) reduces plasma F2 isoprostane and increases potential antioxidant (PAO) levels.
3. To assess the tolerability of Cerefolin® NAC
4. To explore the effects of Cerefolin® NAC on a 6-month change in: (a)global and specific cognitive domains in a standardized neuropsychological test battery,(b) quality of life as measured by SF-36, (c)instrumental and basic activities of daily living, (d)MADRS; and (e)performance-based physical function.
5. To explore if a change in homocysteine level is related to a change in the plasma glutathione, hs-CRP, IL-6, TNF-α, F2-isoprostane, and PAO levels and to a change in the ratio of Aβ42 to Aβ40.
6. To explore the effects of MS AG2756, APOE and MFTHR on the relationship examined in Secondary Objective #5.
7. To explore the relationship of B12 status and status to cognition

NOTE: For individuals successfully completing the 6-month blinded phase, there is an 12-month open-label extension of Cerefolin NAC + multivitamin. The primary purpose of the exploratory, open-label extension phase of the CERE-001 study is to systematically collect long-term safety data on CEREFOLIN NAC usage over an additional 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 60;
* Memory complaints as defined by two questions:

  1. "Do The subject think your have memory problems?"; and,
  2. "Has there been a decline in your memory over the last 10 years?"
* Fluency in English;
* Ability to ingest oral medications; and,
* Willing to replace current vitamin intake with a standardized multivitamin provided for the study.

Exclusion Criteria:

* Clinical stroke or Parkinson's disease;
* Taking FDA approved drug for symptomatic treatment of Alzheimer's disease (Aricept, Razadyne, Exelon, and/or Namenda);
* History of significant renal insufficiency (creatinine ≥1.5);
* History of renal stones or peptic ulcer disease;
* Use of vitamin supplements containing more than 400mcg of folic acid per day within 2 months of Screen Visit;
* As determined by the study physician, clinically significant serum folate and vitamin B12 deficiency on screening blood tests that would require further clinical evaluation and treatment
* As determined by the study physician, clinically significant medical conditions, physical exam findings or abnormal blood tests at screening that would require further clinical evaluation and treatment
* B12 injections 6 months prior to the Screen Visit;
* Confirmed clinical diagnosis of Mild Cognitive Impairment (MCI), vascular dementia or Alzheimer's Disease (AD); and,
* Known hypersensitivity to L-methylfolate, methyl-cobalamin or N-acetylcysteine.
* Use of any other investigational agent used during the 30 days prior to Screening.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj C Shah, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Alzheimer's Disease Center, Chicago, Illinois, United States

REFERENCES:
- See also: Rush Alzheimer's Disease Center — http://www.rush.edu/radc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and September 2009, persons expressing study interest at community presentations or at the Rush Memory Clinic were contacted. Of 524 persons expressing interest, 400 were excluded before consenting for having excluding clinical diagnoses(227), participation refusal (119), and other exclusions medication (54).
Pre-assignment Details: Consented participants underwent a screening evaluation to ensure inclusion criteria were met prior to study treatment assignment and one month run-in treatment with a multivitamin only. Of 124 consented individuals, 20 discontinued prior to randomization due to new medical conditions (9), declining participation (5), and for other reasons (6).
Groups:
- Cerefolin NAC + Multivitamin: On Cerefolin NAC and open-label multivitamin supplement
  Cerefolin NAC (a medical food) : Cerefolin NAC one tablet each day
- Cerefolin NAC Placebo + Multivitamin: On placebo and open label multivitamin supplement
  Cerefolin NAC placebo : Placebo tablet once a day
Period: Overall Study
Arm/Group | Cerefolin NAC + Multivitamin | Cerefolin NAC Placebo + Multivitamin
Started | 51 | 53
Completed | 43 (All participants started (51) were included in primary analyses.) | 49 (All participants started (53) were included in primary analyses.)
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cerefolin NAC + Multivitamin | Cerefolin NAC Placebo + Multivitamin | Total
Number analyzed (Participants) | 51 | 53 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 80.9 (6.6) | 79.4 (8.7) | 80.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 88
  Male | 5 | 11 | 16
Region of Enrollment [Number; unit: participants]
  United States | 51 | 53 | 104
Education Level [Mean (Standard Deviation); unit: years] | 15 (3) | 15 (3) | 15 (3)
total plasma homocysteine [Geometric Mean (Standard Deviation); unit: micromol/L] | 8.35 (1.32) | 8.10 (1.33) | 8.22 (1.33)
glutathione [Geometric Mean (Standard Deviation); unit: micromol/L] | 4.01 (1.67) | 4.02 (1.59) | 4.02 (1.63)
ratio of amyloid beta 1-42 to 1-40 [Geometric Mean (Standard Deviation); unit: pmol/L:pmol/L] | 0.027 (1.73) | 0.034 (1.81) | 0.031 (1.77)
highly sensitive c-Reactive Protein [Geometric Mean (Standard Deviation); unit: mg/mL] | 0.20 (18.93) | 0.23 (22.37) | 0.22 (20.68)
tumor necrosis factor alpha [Geometric Mean (Standard Deviation); unit: pg/mL] | 1.45 (1.61) | 1.37 (1.53) | 1.41 (1.57)
interleukin-6 [Geometric Mean (Standard Deviation); unit: pg/mL] | 2.12 (1.98) | 2.12 (2.35) | 2.12 (2.17)
malondialdehyde [Geometric Mean (Standard Deviation); unit: micromol/L] | 0.90 (1.67) | 0.93 (1.75) | 0.92 (1.71)
potential anti-oxidant (PAO) [Geometric Mean (Standard Deviation); unit: micromol/L] — Potential anti-oxidant (PAO) measures the antioxidant capacity of a serum sample to reduce cupric ions from Cu++ to Cu+.
  micromol/L | 979 (2) | 1016 (2) | 997 (2)

OUTCOME MEASURES:

1. Primary Outcome: Six Month Blood Levels of Homocysteine, Glutathione, and the Ratio of Aβ42 to Aβ40 (as a Percent of Baseline Levels) After Daily Intake of Cerefolin NAC Plus a Multivitamin Versus a Multivitamin Only
Description: Primary outcome markers were plasma homocysteine (tHcy), glutathione, and the ratio of amyloid proteins, Aβ42 and Aβ40. Plasma tHcy and glutathione were assayed using a high performance liquid chromatography (HPLC) with fluorescence detection method. Enzyme-linked immunosorbent assays (ELISA) were used for Aβ42 (Wako Chemicals USA, Inc., Richmond, VA) and Aβ40 (Invitrogen Corporation, Canarillo, CA) detection. Primary analyses utilized Last Observation Carried Forward (LOCF) to assess the primary biomarker level at 6 months versus baseline. Six month levels in biomarker outcomes were compared using t-tests of the logarithmically transformed values and the antilogarithm was applied to the SDs obtain 95% confidence intervals (95% CIs). A significant difference between treatments was needed for at least one of the primary outcome variables (tHcy, glutathione, or the Aβ42 to Aβ40 ratio) to declare the study positive.
Time Frame: 6 months
Population: The Intent-to-Treat (ITT) cohort included randomized subjects taking at least one study treatment dose. Primary analyses utilized Last Observation Carried Forward (LOCF) to assess 6 month levels in the primary biomarkers. 2-sided, t-test p-value for group differences was only significant (<0.05) for 6-month homocysteine level.
Measure: Mean (95% Confidence Interval); unit: percent of baseline level
Groups:
- Cerefolin NAC + Multivitamin: On Cerefolin NAC and open-label multivitamin supplement
- Cerefolin NAC Placebo + Multivitamin: On placebo and open-label multivitamin supplement
Arm/Group | Cerefolin NAC + Multivitamin | Cerefolin NAC Placebo + Multivitamin
Number analyzed (Participants) | 51 | 53
percent of baseline level
  6-Month Homocysteine Level | 71 [66 to 77] | 101 [96 to 107]
  6-Month Glutathione Level | 115 [101 to 129] | 101 [85 to 117]
  6-Month AB42/AB40 Ratio | 101 [92 to 110] | 104 [97 to 108]

2. Secondary Outcome: Tolerability of Cerefolin NAC and a Multivitamin Versus a Multivitamin Only
Description: Mean study product compliance was measured as the actual number of study product tablets taken as a percent of the maximum study product tablets that could have been taken during the intervention period.
Time Frame: 6 months
Population: All participants in Intent-to-Treat cohort were included.
Measure: Mean (Standard Error); unit: percent of study drug taken
Arm/Group | Cerefolin NAC + Multivitamin | Cerefolin NAC Placebo + Multivitamin
Number analyzed (Participants) | 51 | 53
percent of study drug taken | 88 (15) | 88 (21)

3. Secondary Outcome: Six Month Levels of Inflammation and Oxidative Stress Markers(as a Percent of Baseline Levels) After Daily Treatment With Cerefolin NAC and a Multivitamin or a Multivitamin Only
Description: Outcome measures were 6-month levels of highly sensitive c-reactive protein (hs-CRP), tumor necrosis factor alpha (TNF-alpha), interleukin-6 (IL-6), malondialdehyde, and potential anti-oxidant (PAO)in blood samples as a percent of baseline value.
Time Frame: 6 months
Population: All participants in Intent-to-Treat were included with last observation carried forward.
Measure: Mean (95% Confidence Interval); unit: percent of baseline level
Arm/Group | Cerefolin NAC + Multivitamin | Cerefolin NAC Placebo + Multivitamin
Number analyzed (Participants) | 51 | 53
percent of baseline level
  6-month hs-CRP Level | 110 [51 to 238] | 111 [53 to 234]
  6-month TNF-alpha Level | 99 [93 to 106] | 108 [98 to 118]
  6-month IL-6 Level | 114 [97 to 134] | 105 [88 to 125]
  6-month Malondialdehyde Level | 93 [83 to 104] | 90 [79 to 102]
  6-month PAO Level | 109 [96 to 123] | 115 [100 to 131]

ADVERSE EVENTS:
Arm/Group | Cerefolin NAC + Multivitamin | Cerefolin NAC Placebo + Multivitamin
Serious Adverse Events (participants affected / at risk) | 11/51 | 8/53
Other Adverse Events (participants affected / at risk) | 30/51 | 28/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cerefolin NAC + Multivitamin (N=51) | Cerefolin NAC Placebo + Multivitamin (N=53)
Cardiac disorders (Cardiac disorders) | 3 (3) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 0 (0)
General Disorders (General disorders) | 2 (2) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 3 (3) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cerefolin NAC + Multivitamin (N=51) | Cerefolin NAC Placebo + Multivitamin (N=53)
Cardiac disorders (Cardiac disorders) | 1 (1) | 2 (3)
Eye disorders (Eye disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (6) | 3 (4)
General disorders (General disorders) | 4 (4) | 5 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (7)
Nervous system disorders (Nervous system disorders) | 2 (2) | 5 (5)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)

LIMITATIONS AND CAVEATS:
No limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No